CLINICAL TRIAL: NCT02603991
Title: Prospective Cohort Study on the Efficacy of Vagus Nerve Stimulation for Children and Adolescents With Epilepsy(PVNS-CAE)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Pins Medical Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: PINS-015
Record Dates: First submitted 2015-11-09; First posted 2015-11-13 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Epileptic Encephalopathy
Keywords: children and adolescents; Prospective cohort study; vagus nerve stimulation; PINS
MeSH Terms: interventions — Levetiracetam

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: PINS Vagus Nerve Stimulator — The stimulators are implanted in the body,with the stimulation of the IPG
Drug: Levetiracetam — The best anti-epileptic drugs to patients who participate in this study，Levetiracetam，

SUMMARY:
Prospective cohort study on the long-term effectiveness and safety of PINS vagus nerve stimulators for children and adolescent with refractory epilepsy.

DETAILED DESCRIPTION:
Epileptic encephalopathy is very common in children and adolescent with epilepsy, but there is no data in clinical studies.The aim of this study is to evaluate the efficacy of the long-term vagus nerve stimulation for children and adolescent with epilepsy

ELIGIBILITY:
Inclusion Criteria:

1. age 4-18
2. Diagnostic criteria for epilepsia brain disorders
3. Having tried appropriate anti-epileptic drugs (AEDs) more than 1 year and zt least 6 seizures per month
4. patients or his(her) families could understand this method and sign the informed consent
5. Patients with good compliance and could complete postoperative follow-up

Exclusion Criteria:

1. the vagus nerve lesion and damage
2. patients with progressive neurological diseases, cardiopulmonary anomaly, respiratory system diseases,digestive system diseases
3. patients'mental state is not stable，
4. patients with or anesthesia contraindications,such as long-term use of anticoagulation antiplatelet drugs etc.
5. patients have or need other implantable devices, such as pacemakers,defibrillators, cochlear and spinal nerve root stimulator.
6. patients due to their own reasons for the need for nuclear magnetic resonance imaging in the future clinical trials
7. patients have participated in other clinical trials.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients at age 4-18; diagnostic criteria for epilepsia brain disorders; having tried appropriate anti-epileptic drugs (AEDs) more than 1 year and at least 6 seizures per month; patients or his(her) familys could understand this method and sign the informed consent; Patients with good compliance and could complete postoperative follow-up；without the vagus nerve lesion and damagement, progressive neurological diseases, cardiopulmonary anomaly, respiratory system diseases, digestive system diseases
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-01 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
The change of the score in Quality of Life in Children with Epilepsy | QOLCE Scores at 3,6,9,12,18, 24 month of stimulation

SECONDARY OUTCOMES:
Respondent rate | Respondent rate at 3,6,9,12,24 month
seizure free rate | seizure free rate at 3,6,9,12, 24 month
complication | complication at 3,6,9,12, 24 month

CONTACTS AND LOCATIONS:
Overall Officials: Jianguo Zhang, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China